CLINICAL TRIAL: NCT00024596
Title: Family Heart Study - Subclinical Atherosclerosis Network (FHS-SCAN)
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michael Province, Professor of Genetics and Biostatistics, Washington University School of Medicine
Other Study IDs: 985; R01HL088215 (NIH)
Record Dates: First submitted 2001-09-21; First posted 2001-09-21 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Atherosclerosis; Coronary Arteriosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Atherosclerosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Stored DNA, lymphoblasts

GROUPS / COHORTS (2):
- Caucasian Families: Largest 3-generational Caucasian Families from Family Heart Study (Classic) with average family size of 10 N=2767 Subjects from 512 families. Approximately half are random sample families from FamHS-Classic, and half are high-familial CHD risk families from FamHS-Classic. 4 Field sites were Raleigh-Durham North Carolina; Minneapolis, MN; Framingham MA; and Salt Lake City, UT.
- African-American Families: 622 subjects from 2-3 generational 212 African-American families originally recruited from the HyperGEN study in Birmingham AL. These are hypertension enriched families.

SUMMARY:
To determine familial and non-familial causes for susceptibility to atherosclerosis and the inflammatory response.

DETAILED DESCRIPTION:
BACKGROUND:

Atherosclerotic cardiovascular disease, along with its related health expenditures, mortality, and morbidity, remains among the most significant health-related conditions in the United States and other developed countries. The substantial resources that have been expended to investigate this problem have led to significant scientific advances in the basic biology, clinical management, epidemiology, and public health intervention approaches. Despite these real advances, there remains much more to be done in terms of understanding the basic biological and social processes, treatment, and public health programs.

Just as earlier research was effective in identifying a variety of epidemiologic risk factors for cardiovascular disease, recent advances make it possible to bring to bear a variety of new and powerful tools to detailed study of the basic processes involved in atherogenesis. Application of these tools, in combination with synthesis of prior basic and epidemiologic results, provides a powerful approach that is more model-driven than many previous studies.

DESIGN NARRATIVE:

The Subclinical Atherosclerosis Network is a multicenter study of the genetic epidemiology of coronary and aortic calcification and of inflammatory markers. It examines two areas of great interest in contemporary vascular medicine, namely vascular calcification and inflammation in approximately 3000 persons who have been recruited to the Family Heart Study, with additional persons of African American descent contributed by the HyperGEN Study. Considerable data, including a large number of genotypes, have been collected in the Family Heart Study. The subjects will be brought back for additional data collection, including the measurement of inflammatory markers and coronary and aortic calcification by computed tomography (CT).

The network will quantify coronary and aortic artery calcium volume in 441 selected, informative pedigrees ( approximately 3,000 individuals) previously examined and extensively genotyped ( approximately 400 markers spanning the genome) by the NHLBI Family Heart Study, in order to identify genes associated with human atherosclerosis. An additional 275 African American sibships (approximately 600 individuals, also examined and comparably genotyped) will be included to address these study questions in this high-risk population. Assessment of the inter-individual variability in the inflammatory burden and the host response, and the extensive metabolic, behavioral, and environmental data already collected on these pedigrees will provide enhanced phenotypic homogeneity and increased analytic power in assessing the genetic basis of atherosclerosis.

State of the art laboratory and statistical methods will be used to find, localize and characterize the influence of predisposing genes to atherosclerosis and the inflammatory response. Novel genetic analysis methods will be used to address the issues of phenotypic, genetic and population heterogeneity, epistasis, complex interactions among the genetic and environmental risk factors, and to optimize the detection of genomic regions affecting phenotypic susceptibility.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3389 (Actual)
Dates: Start 2001-09; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Carr — Wake Forest University; John Eckfeldt — University of Minnesota; R. Ellison — Boston University; Gerardo Heiss — University of North Carolina; James Hixson — University of Texas; Steven Hunt — University of Utah; Cora Lewis — University of Alabama at Birmingham; James Pankow — University of Minnesota; Michael Province — Washington University School of Medicine; Lynne Wagenknecht — Wake Forest University

REFERENCES:
- [Background] Djousse L, Arnett DK, Carr JJ, Eckfeldt JH, Hopkins PN, Province MA, Ellison RC; Investigators of the NHLBI FHS. Dietary linolenic acid is inversely associated with calcified atherosclerotic plaque in the coronary arteries: the National Heart, Lung, and Blood Institute Family Heart Study. Circulation. 2005 Jun 7;111(22):2921-6. doi: 10.1161/CIRCULATIONAHA.104.489534. Epub 2005 May 31. PMID 15927976
- [Background] Ellison RC, Zhang Y, Wagenknecht LE, Eckfeldt JH, Hopkins PN, Pankow JS, Djousse L, Carr JJ. Relation of the metabolic syndrome to calcified atherosclerotic plaque in the coronary arteries and aorta. Am J Cardiol. 2005 May 15;95(10):1180-6. doi: 10.1016/j.amjcard.2005.01.046. PMID 15877990